CLINICAL TRIAL: NCT06034249
Title: The Effect of Mindfulness-Based VR on Depression, Sleep and Quality of Life Among Family Caregivers of People With Dementia
Brief Title: Mindfulness-Based VR for Family Caregivers of People With Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University (Other)
Collaborators: National Science and Technology Council (U.S. Federal Agency)
Responsible Party: Principal Investigator, Megan F. Liu, Associate Professor, Taipei Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 20230816
Record Dates: First submitted 2023-09-05; First posted 2023-09-13 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Caregivers of People With Dementia; Quality of Life
Keywords: Virtual Reality; Depression; Sleep Quality
MeSH Terms: conditions — Depression; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: A randomized controlled trial (RCT) design was used. Participants will be ask to attend the six-week course encompassed various mindfulness practices, including breathing observation, body scanning, mindful yoga, mindful walking, holistic meditation, and non-selective awareness practices. The control group will only be given the mindfulness-based audio files for six weeks.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group: Mindfulness-Based VR group (Experimental): Participants will be ask to attend the six-week course encompassed various mindfulness practices, including breathing observation, body scanning, mindful yoga, mindful walking, holistic meditation, and non-selective awareness practices.
  Interventions: Behavioral: Mindfulness-Based VR
- Control Group: Mindfulness-based Audio Files (Placebo Comparator): The control group will only be given the mindfulness-based audio files for six weeks.
  Interventions: Behavioral: Audio

INTERVENTIONS:
Behavioral: Mindfulness-Based VR — Participants will be ask to attend the six-week course encompassed various mindfulness practices, including breathing observation, body scanning, mindful yoga, mindful walking, holistic meditation, and non-selective awareness practices.
  Arms: Experimental Group: Mindfulness-Based VR group
Behavioral: Audio — The mindfulness-based audio files for six weeks.
  Arms: Control Group: Mindfulness-based Audio Files

SUMMARY:
The goal of this clinical trial is to explore the effectiveness of mindfulness-based VR could enhance depression, sleep quality, and overall quality of life for family caregivers providing care for people with dementia.

Participants will be ask to attend the six-week course encompassed various mindfulness practices, including breathing observation, body scanning, mindful yoga, mindful walking, holistic meditation, and non-selective awareness practices. The control group will only be given the mindfulness-based audio files for six weeks.

DETAILED DESCRIPTION:
The inclusion criteria for participants were as follows: (1) being a family caregiver responsible for caring for a family member diagnosed with dementia by a medical institution, (2) having the ability to communicate in Mandarin or Taiwanese, and (3) providing informed consent to participate in the study by signing the consent form. Individuals with visual and auditory impairments were excluded from the study.

Outcome measure: basic characteristics of participants; The Center for Epidemiologic Studies Depression Scale; Questionnaire of Taiwan's World Health Organization Quality of Life Brief Version.

ELIGIBILITY:
Inclusion Criteria:

1. being a family caregiver responsible for caring for a family member diagnosed with dementia by a medical institution,
2. having the ability to communicate in Mandarin or Taiwanese, and
3. providing informed consent to participate in the study by signing the consent form.

Exclusion Criteria:

Visual and auditory impairments were excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2022-08-23 (Actual); Primary Completion 2022-11-21 (Actual); Study Completion 2023-06-06 (Actual)

PRIMARY OUTCOMES:
Depression | Baseline and six-week
  The Center for Epidemiologic Studies Depression Scale (CES-D) The minimum value= 0, maximum value= 60, higher score mean higher frequency of depressive symptoms.

SECONDARY OUTCOMES:
Sleep | Baseline and six-week
  Chinese Pittsburgh Sleep Quality Index (CPSQI) The minimum value= 0, maximum value= 21, higher score mean worse sleep quality.
QoL | Baseline and six-week
  Questionnaire of Taiwan's World Health Organization Quality of Life Brief Version The minimum value= 4, maximum value= 20, higher score mean better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Megan F Liu, PhD, Principal Investigator — Taipei Medical University
Locations (1):
- Taipei Medical University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
No plan to make individual participant data (IPD) available to other researchers.